CLINICAL TRIAL: NCT02481102
Title: EASYER (EpiAccess SYstem Registry) - A Post Market Observational Registry
Brief Title: EASYER (EpiAccess SYstem Registry) A Post Market Observational Registry
Acronym: EASYER
Status: Completed | Type: Observational
Sponsor: EpiEP, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: QT-0020
Record Dates: First submitted 2015-06-18; First posted 2015-06-25 (Estimated); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Arrhythmias, Cardiac
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Days
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of the Registry is to provide post market clinical outcome and potential health economics data and confirm the continued safety of the EpiAccess system.

DETAILED DESCRIPTION:
The Registry will be a prospective non-randomized single-arm trial of up to 150 patients enrolled in up to ten (10) centers in the United States. The overall duration of the registry is estimated to be 18 months per site. For the patients the registry duration will be from the time of procedure until discharge from the hospital, estimated to be approximately four (4) days.

Prior to enrollment, patients will be evaluated on the basis of the latest available data to establish eligibility. Eligible patients will be considered enrolled in the registry after written informed consent is obtained.

As EpiAccess is only used for the access portion of the procedure, the safety performance and effectiveness endpoints are acute from the time of needle insertion until pericardial sac access is achieved. Follow up clinical examinations will be performed according to institutional standard of care. No special tests are required for this device.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 years of age or older
* Pericardial access is clinically indicated
* Patient is willing and able to provide written informed consent

Exclusion Criteria:

* Patients who have any condition which contraindicates pericardial access or who have any condition specified in the Contraindications section of the Instructions for Use. This includes:
* Previous cardiac surgery or myocardial infarctions resulting in pericardial fibrosis
* Congenital absence of a pericardium
* Absence of a free epicardial space
* Patients with active infection
* History of chronic pericarditis
* Patient requiring anti-arrhythmic drug therapy for the treatment of ventricular arrhythmia
* Patient not in normal sinus rhythm
* Presence of thrombus in the left atrium
* Coagulopathy
* Known allergy to contrast media

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are clinically indicated for a procedure requiring pericardial access are eligible for the study.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2015-06-30 (Actual); Primary Completion 2021-02-09 (Actual); Study Completion 2021-02-09 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as Measure of Safety | Up to 4 days post procedure (or until time of discharge)
  Number of Participants with Adverse Events as Measure of Safety

SECONDARY OUTCOMES:
Health Economics | Up to 4 days post procedure (or until time of discharge)
  Number of Participants with Extended Hospital Stay as a Measure of Health Economic Value

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Natale, MD, Principal Investigator — Texas Cardiac Arrhythmia Research Foundation; Vivek Reddy, MD, Principal Investigator — Icahn School of Medicine, Mount Sinai Hospital
Locations (3):
- United States (3):
  - Vivek Reddy, New York, New York
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Texas Cardiac Arrhythmia, Austin, Texas

IPD SHARING:
Plan to Share IPD: No